CLINICAL TRIAL: NCT02521363
Title: Pilot Trial of an Implantable Microdevice for In Vivo Drug Sensitivity Testing in Patients With Early Stage, HER2-Positive or Triple Negative Breast Cancer
Brief Title: Implantable Microdevice for In Vivo Drug Sensitivity Testing in Patients With Early Stage, HER2-Positive or Triple Negative Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15-127
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Results first posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
Keywords: Implantable Microdevice; In Vivo Drug Sensitivity Testing; HER2-Positive; Triple Negative; 15-127
MeSH Terms: conditions — Breast Neoplasms | interventions — Anthracyclines

ARMS (2):
- Upfront Breast Surgery (Experimental): Patients will have the microdevice implanted prior to breast surgery, in the absence of neoadjuvant chemotherapy
  Interventions: Device: KIBUR MICRODEVICE
- Neoadjuvant Therapy (Experimental): Patients will have the device placed and retrieved on a core biopsy the following day, then receive neoadjuvant chemotherapy prior to definitive breast surgery.
  Interventions: Device: KIBUR MICRODEVICE; Drug: anthracycline and taxane based chemotherapy

INTERVENTIONS:
Device: KIBUR MICRODEVICE — This device contains 16 reservoirs, each with a unique single agent or drug combination in microdose amounts of less than one millionth of a systemic patient dose. The device is implanted directly into the tumor during a biopsy procedure, and remains in situ for ~24 hours.
Drug: anthracycline and taxane based chemotherapy — Conventional, standard of care neoadjuvant chemotherapy delivered irrespective of device readout
  Arms: Neoadjuvant Therapy

SUMMARY:
The purpose of this study is to test the safety and feasibility of placing and removing a small device that contains anti-cancer drugs in a breast tumor of patients who plan on having breast surgery without treatment prior or patients who plan on receiving standard preoperative chemotherapy prior to their breast surgery. This device may be able to predict what types of treatment work best against an individual's breast cancer. With this device, the investigators hope to be able to personalize treatment choices based on an individual's type of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed invasive breast cancer that is: Triple negative (ER<10%, PR<10%, and HER2 0/1+ or 2+/FISH not amplified)
* Tumor size 2cm or greater; N any; M0
* Tumor size 1cm or greater; N any; M0 (Cohort 1)
* Tumor size 2cm or greater; N any; M0 (Cohort 2)
* Candidate for curative breast cancer surgery (Cohort 1 or 2)
* Candidate for neoadjuvant chemotherapy with a standard of care, anthracycline-based regimen (Cohort 2 preferred over Cohort 1)
* Age >18 years of age
* ECOG performance status of ≤2
* Serum or urine pregnancy test negative within 2 weeks for women of childbearing potential.
* Willing and able to provide informed consent

Exclusion Criteria:

* Prior treatment including surgery, chemotherapy or radiation therapy for the current primary breast cancer.
* Severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational device administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Traina, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan-Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center at Mercy Medical Center, Rockville Centre, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Upfront Breast Surgery | Neoadjuvant Therapy
Started | 4 | 7
Completed | 3 | 5
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Upfront Breast Surgery | Neoadjuvant Therapy | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Full Range); unit: years] | 55.5 [52 to 60] | 43.9 [32 to 54] | 48 [32 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4 | 7 | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Implantable Devices
Description: If we are able to collect data from at least 6 out of the 12 patients, we will deem this study feasible to conduct in a larger cohort of patients.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Upfront Breast Surgery | Neoadjuvant Therapy
Number analyzed (Participants) | 4 | 7
Participants
  Participants with implantable devices | 3 | 5
  Not evaluable | 1 | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Upfront Breast Surgery | Neoadjuvant Therapy
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 0/4 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-22): https://cdn.clinicaltrials.gov/large-docs/63/NCT02521363/Prot_SAP_000.pdf